CLINICAL TRIAL: NCT03231605
Title: Comparative Immunogenicity Study of Two Live Attenuated Hepatitis A Vaccines
Brief Title: Comparative Immunogenicity Study of Two Hepatitis A Vaccines
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Shaanxi Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91110000100010062X
Record Dates: First submitted 2017-07-20; First posted 2017-07-27 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 is experimental group which used the Hepatitis A Vaccine product by Changchun Institute of Biological Co.,Ltd
  Interventions: Biological: Hepatitis A Vaccine
- Group 2 (Active Comparator): Group 2 is control group which used the Hepatitis A Vaccine product by Changchun Changsheng Life Sciences Limited
  Interventions: Biological: Hepatitis A Vaccine

INTERVENTIONS:
Biological: Hepatitis A Vaccine — Vaccinating two Hepatitis A Vaccines separately in 18-24 months Children based on the grouping result .

SUMMARY:
Hepatitis A is the most prevalent hepatitis which account for approximately 45% . The susceptible population is Children and adolescence, also the morbidity in adult presented rising trend in recent years. Therefore, vaccination of Hepatitis A Vaccine play an important role in National Immunisation Program(China). The aim of this experiment is to verify the effects of experimental group non-inferior than control group. The experiment methods is compared the difference of seroconversion rate and Antibody geometric mean titer (GMT)between experimental and control Hepatitis A Vaccines. In addition, evaluating the safety of two Hepatitis A Vaccines in 18-24 months Chinese Children.

ELIGIBILITY:
Inclusion Criteria:

* The healthy children in mental and physical aged between 18-24 months, and the guardians agree and fully understand the protocol.
* No Hepatitis A disease and contraindication of vaccination
* No history of Hepatitis A Vaccine
* The subjects can follow the requirements of experiment project.
* Do not vaccinate other vaccine in one months.
* Axillary's temperature≤37℃

Exclusion Criteria:

* Having severe diseases.
* Allergy to the components in Vaccine
* Immune abnormalities
* The people who do not agree with the Inclusion Criteria
* Have a serious chronic disease
* Any conditions which researcher think will influence the results or the subjects.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-12-29 (Estimated)

PRIMARY OUTCOMES:
To verify the protection rate and antibody quantity of experimental vaccine non-inferior than control vaccine. | 35-42 days
  Collecting serum of subjects before, after vaccination immediately and after 35-42 days, and testing the quantity of antibody. Compared the difference of antibody quantity between two types Hepatitis A Vaccine and the Multiple of antibody based on the time.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 month
  Observation 30 minutes after vaccination and give guardians feedback forms to record untoward effects, collecting the forms after 1 month when the subjects conduct the third time blood collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Provincial Center for Disease Control and Prevention, Yuncheng, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
Based on the literature public progress.

REFERENCES:
- See also: The reference 6 — https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/Vaccines/UCM164319.pdf
- See also: The reference 8 — http://med.wanfangdata.com.cn/Paper/Detail?id=PeriodicalPaper_zgswzpxzz200909021
- See also: The reference 9 — http://www.wenkuxiazai.com/doc/c36ab52c58fb770bf78a5529.html